CLINICAL TRIAL: NCT01552902
Title: A Phase 4, Randomized, Double-blind, Multicenter, Parallel-group, Active-controlled, Forced-dose Titration, Safety and Efficacy Study of SPD489 (VYVANSE®) Compared With OROS-MPH (CONCERTA®) With a Placebo Reference Arm, in Adolescents Aged 13-17 Years With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: Effectiveness of Vyvanse Compared to Concerta in Adolescents With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-406; 2011-005452-34 (EudraCT Number)
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lisdexamfetamine dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine dimesylate
- Methylphenidate Hydrochloride (Active Comparator)
  Interventions: Drug: Methylphenidate Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — Daily oral dosing in the AM ranging from 30- 70 mg. 4 week forced dose titration, 2 week dose maintenance
  Other Names: SPD489, Vyvanse, LDX
  Arms: Lisdexamfetamine dimesylate
Drug: Methylphenidate Hydrochloride — Daily oral dosing in the AM ranging from 18-72 mg. 4 week force dose titration, 2 week dose maintenance
  Other Names: Concerta, OROS-MPH
  Arms: Methylphenidate Hydrochloride
Drug: Placebo — Daily oral dosing in the AM for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine effectiveness of Vyvanse compared to Concerta in adolescents with Attention-deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 13-17 years of age, inclusive, at the time of consent.
* Subject must weigh more than 79.5lb.
* The parent/LAR must be available at approximately 7:00AM (±2 hours) to dispense the dose of investigational product for the study duration.
* Subject, who is a female, must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test and a negative urine pregnancy test and agree to comply with any applicable contraceptive requirements of the protocol.
* Subject has an ADHD-RS-IV total score ≥28.
* Subject is able to swallow a capsule.
* Subject does not have hypertension and has a resting sitting blood pressure less than or equal to 135/85mmHg.

Exclusion Criteria

* Subject has a current, controlled (with medications prohibited in this study) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any significant comorbid Axis II disorder or significant Axis I disorder (such as post traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, depressive or anxiety disorder.
* Diagnosis of conduct disorder. Oppositional defiant disorder is not exclusionary.
* Subject is considered a suicide risk, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded.
* Subject is underweight or overweight.
* Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition. Mild, stable asthma is not exclusionary.
* Subject has a history of seizures (other than infantile febrile seizures), a chronic or current tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
* Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place him/her at increased vulnerability to the sympathomimetic effects of a stimulant medication.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subject has any clinically significant ECG or clinically significant laboratory abnormality.
* Subject has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone (TSH) and thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
* Subject has a documented allergy, hypersensitivity, or intolerance to MPH or to any excipients in the reference product.
* Subject has failed to fully respond to an adequate course(s) (dose and duration) of MPH or amphetamine therapy.
* Subject has a history of suspected substance abuse or dependence disorder (excluding nicotine). Subjects with a lifetime history of amphetamine, cocaine, or other stimulant abuse and/or dependence will be excluded.
* Subject has a positive urine drug result.
* Subject has previously participated in this study or another clinical study involving SPD489/NRP104.
* Subject has glaucoma.
* Subject is required to take or anticipates the need to take medications that have CNS effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
* Subject is female and is pregnant or lactating.
* Subject is well controlled on his/her current ADHD medication.
* Subject has a pre-existing severe gastrointestinal tract narrowing.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 549 (Actual)
Dates: Start 2012-04-03 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2014-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (95):
- United States (81):
  - Harmonex Neuroscience Research, Inc., Dothan, Alabama
  - Center for Advanced Improvement, Tucson, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Shanti Clinical Trials, Colton, California
  - Sun Valley Research Center, Imperial, California
  - Synergy Clinical Research Center, National City, California
  - Pacific Sleep Medicine, A Medical Corporation, Oceanside, California
  - Neuropsychiatric Research Center for Orange County, Orange, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - PCSD - Feighner Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Elite Clinical Trials, Wildomar, California
  - IMMUNOe International Research Center, Centennial, Colorado
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Amedica Research Institute, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Sarkis Clinical Trials, Lake City, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Prevention & Strengthening Solutions, Inc., Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Atlanta Institute of Medicine & Research, Inc, Atlanta, Georgia
  - Clinical Research Center, University of Illinois at Chicago, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - Pedia Research, LLC, Newburgh, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Louisiana Resarch Associates, Inc., New Orleans, Louisiana
  - Marc Hertzman, MD, PC, Rockville, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, PC, Sterling Heights, Michigan
  - Behavioral Medical Center - Troy, Troy, Michigan
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - Psychiatric Care & Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - University of Nebraska Medical Center Dept Of Psychiatry, Omaha, Nebraska
  - Center for Psychiatry & Behavioral Medicine, Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Brain Resource Center, New York, New York
  - Mount Sinai School of Medicine/Dept of Psychiaatry, New York, New York
  - Duke University medical Center/ Duke ADHD Program, Durham, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - University of Cincinnati College of Medicine/UCPC, Cincinnati, Ohio
  - The Ohio State University Nisonger Center, Columbus, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Center for Clinical Investigations Inc, Portland, Oregon
  - Summit Research Network, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - University Services, West Chester, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Rainbow Research, Inc., Barnwell, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Research Across America/Psychiatric Medical Associates, Dallas, Texas
  - Bayou City Research, Houston, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Ericksen Research and Development - Westside Medical, Clinton, Utah
  - University of Virginia Child and Family Psychiatry Clinic, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Thereapeutic Resource, Kirkland, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington
  - Rockwood Clinic, P.S., Spokane, Washington
- Canada (2):
  - True North Clinical Research, Kentville, Nova Scotia
  - The Kids Clinic, Whitby, Ontario
- Germany (6):
  - Schwerpunktpraxis fur Entwicklung und Lernen, Bamberg
  - Klinik Fur Kinder- und Jugendpsychiatrie, Psychosomatik und Psychotherapie, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Kinderarztpraxis Dr. Kaiser und Dr. MarineBe, Hamburg
  - Zentralinstitut fur Seelische Gesundheit, Mannheim
  - Medizinisches Studienzentrum Wurzburg, Würzburg
- Hungary (4):
  - Vadaskert Gyermekpszichiatriai Korhaz es Szakambulancia, Budapest
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Pecsi Megyei Jogu varos Egyesitett Egeszsegugyi Intezmenyek, Pécs
  - Szegedi Tudomanyegyetem, Szeged
- Sweden (2):
  - Gillbergcentrum, Gothenburg
  - PRIMA Barn-och Vuxenpsykiatri Jarva, Spånga

REFERENCES:
- [Derived] Newcorn JH, Nagy P, Childress AC, Frick G, Yan B, Pliszka S. Randomized, Double-Blind, Placebo-Controlled Acute Comparator Trials of Lisdexamfetamine and Extended-Release Methylphenidate in Adolescents With Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2017 Nov;31(11):999-1014. doi: 10.1007/s40263-017-0468-2. PMID 28980198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 77 sites in the United States, Canada, and Europe.
Pre-assignment Details: Of the 778 screened participants, 229 were screen failures and 549 were randomized to treatment. A total of 547 participants were treated and the reasons for 2 'randomized but not treated' participants included withdrawal by 1 participant in the Methylphenidate group and 1 participant with a protocol violation in the Lisdexamfetamine group.
Groups:
- Placebo: 2 placebo over encapsulated capsules once daily orally for 6 weeks.
- Lisdexamfetamine Dimesylate: Lisdexamfetamine dimesylate (LDX, Vyvanse®, SPD489) 30 to 70 milligram (mg) over encapsulated capsule once daily orally along with placebo over encapsulated capsule for 4 weeks (forced dose titration), followed by LDX 70 mg over encapsulated capsule once daily orally along with placebo over encapsulated capsule for 2 weeks (dose maintenance).
- Methylphenidate: Methylphenidate (Concerta, Osmotic controlled oral release delivery system-methylphenidate [OROS-MPH]) 18 to 72 mg over encapsulated capsule once daily orally along with placebo over encapsulated capsule (no placebo administered when methylphenidate 72 mg [2*36 mg capsules] was administered) for 4 weeks (forced dose titration), followed by methylphenidate 72 mg (2*36 mg capsules) over encapsulated capsule once daily orally for 2 weeks (dose maintenance).
Period: Overall Study
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Started | 110 | 218 | 219
Completed | 97 | 181 | 186
Not Completed | 13 | 37 | 33
Not completed — Adverse Event | 1 | 15 | 14
Not completed — Protocol Violation | 3 | 3 | 3
Not completed — Lack of Efficacy | 4 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 9 | 6
Not completed — Lost to Follow-up | 1 | 3 | 6
Not completed — Other | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Safety set consisted of all participants in the Randomized set (all screened participants for whom a randomization number was generated) who took at least 1 dose of investigational product.
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine dimesylate (LDX, Vyvanse®, SPD489) 30 to 70 mg over encapsulated capsule once daily orally along with placebo over encapsulated capsule for 4 weeks (forced dose titration), followed by LDX 70 mg over encapsulated capsule once daily orally along with placebo over encapsulated capsule for 2 weeks (dose maintenance).
- Methylphenidate: Methylphenidate (Concerta, OROS-MPH) 18 to 72 mg over encapsulated capsule once daily orally along with placebo over encapsulated capsule (no placebo administered when methylphenidate 72 mg [2*36 mg capsules] was administered) for 4 weeks (forced dose titration), followed by methylphenidate 72 mg (2*36 mg capsules) over encapsulated capsule once daily orally for 2 weeks (dose maintenance).
- Total: Total of all reporting groups
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate | Total
Number analyzed (Participants) | 110 | 218 | 219 | 547
Age, Categorical [Count of Participants; unit: Participants] — Age was calculated as the difference between date of birth and date of informed consent.
  Participants
    <=18 years | 110 | 218 | 219 | 547
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated as the difference between date of birth and date of informed consent.
  years | 14.7 (1.37) | 14.6 (1.38) | 14.7 (1.42) | 14.7 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 83 | 69 | 186
  Male | 76 | 135 | 150 | 361
Attention-deficit/Hyperactivity Disorder (ADHD) Subtype [Count of Participants; unit: Participants]
  Predominantly Inattentive | 40 | 70 | 71 | 181
  Predominantly Hyperactive/Impulsive | 2 | 2 | 4 | 8
  Combined Subtype | 68 | 146 | 144 | 358
Clinical Global Impressions - Severity of Illness (CGI-S) [Count of Participants; unit: Participants] — The Clinical Global Impressions Scale permits a global evaluation of the participant's severity of illness and improvement over time. The scale includes a severity of illness item and a global improvement item. The investigator performed the CGI-S to rate the severity of a participant's condition on a 7-point scale (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill).
  Participants
    Borderline mentally ill | 1 | 0 | 0 | 1
    Mildly ill | 2 | 4 | 1 | 7
    Moderately ill | 60 | 93 | 115 | 268
    Markedly ill | 41 | 106 | 90 | 237
    Severely ill | 6 | 15 | 13 | 34
Attention-deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Total Score [Mean (Standard Deviation); unit: units on a scale] — The ADHD-RS-IV was developed to measure the behaviors of children with ADHD and is commonly used in clinical studies of ADHD. The ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition-Text Revision (DSM-IV-TR) criteria. Each item was scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54, Higher score = more severe symptoms.
  units on a scale | 36.1 (5.91) | 37.2 (6.46) | 36.9 (6.42) | 36.9 (6.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale, Fourth Edition (ADHD-RS-IV) Total Score at Week 6
Description: The ADHD-RS-IV was developed to measure the behaviors of children with ADHD and is commonly used in clinical studies of ADHD. The ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition-Text Revision (DSM-IV-TR) criteria. Each item was scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54, Higher score = more severe symptoms.
Time Frame: Baseline, Week 6
Population: Full Analysis Set (FAS) was defined as all participants in the Safety set who had at least 1 post-baseline measurement of the ADHD-RS-IV. Not all FAS participants were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Number analyzed (Participants) | 93 | 175 | 181
units on a scale | -17 (1.03) | -25.4 (0.74) | -22.1 (0.73)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Methylphenidate; The least squares mean (LSM), the difference in LSM and its 95% confidence interval (CI), and the p-value were from a mixed effects model for repeated measures that included treatment group, visit, interaction of the treatment group with the visit as factors, baseline score as a covariate, and an adjustment for the interaction of the baseline score with the visit. The model was based on Restricted maximum likelihood (REML) method of estimation and utilized an unstructured covariance; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Difference in LSM = -3.4, 95% CI 2-sided [-5.4 to -1.3]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate; The LSM, the difference in LSM and its 95% CI, and the p-value were from a mixed effects model for repeated measures that included treatment group, visit, interaction of the treatment group with the visit as factors, baseline score as a covariate, and an adjustment for the interaction of the baseline score with the visit. The model was based on REML method of estimation and utilized an unstructured covariance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in LSM = -8.5, 95% CI 2-sided [-11 to -6]
Statistical Analysis 3: Comparison: Placebo vs Methylphenidate; The LSM, the difference in LSM and its 95% CI, and the p-value were from a mixed effects model for repeated measures that includes treatment group, visit, interaction of the treatment group with the visit as factors, baseline score as a covariate, and an adjustment for the interaction of the baseline score with the visit. The model was based on REML method of estimation and utilized an unstructured covariance; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in LSM = -5.1, 95% CI 2-sided [-7.6 to -2.6]

2. Secondary Outcome: Percentage of Participants With an Improvement on Clinical Global Impression - Global Improvement (CGI-I) at Week 6
Description: The Clinical Global Impressions Scale permits a global evaluation of the participant's severity of illness and improvement over time. The scale included a severity of illness item and a global improvement item. The investigator performed the CGI-I to rate the improvement of a participant's ADHD symptoms based on a 7-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse.). Percentage of participants with an improved measurement (response of very much improved and much improved) is reported.
Time Frame: Week 6
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Number analyzed (Participants) | 106 | 210 | 216
percentage of participants | 50 | 81.4 | 71.3

3. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that did not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were events between first dose of double-blind investigational product and up to 3 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 3 days after last dose (last dose at Week 6)
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Number analyzed (Participants) | 110 | 218 | 219
participants
  Participants with TEAEs | 49 | 145 | 129
  Participants with serious TEAEs | 1 | 1 | 1

4. Other Pre Specified Outcome: Change From Baseline in Blood Pressure at Week 6
Time Frame: Baseline, Week 6
Population: Safety set. Not all Safety set participants were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Number analyzed (Participants) | 93 | 175 | 181
millimeter of mercury (mmHg)
  Systolic blood pressure | -1 (9.88) | 1.5 (9.56) | 2.4 (9.97)
  Diastolic blood pressure | -0.1 (8.1) | 3.4 (8.15) | 3.5 (8.59)

5. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Week 6
Time Frame: Baseline, Week 6
Population: Safety set. Not all Safety set participants were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Number analyzed (Participants) | 93 | 175 | 181
Beats per minute | 2.4 (10.81) | 6.7 (12.46) | 8.2 (12.7)

ADVERSE EVENTS:
Time Frame: Baseline up to 3 days after last dose (last dose at Week 6)
Description: AEs occurred during the double-blind evaluation phase were considered as TEAEs if AEs had a start date on or after the first dose of double-blind study drug or a start date before the date of the first dose of double-blind study drug, but increased in severity on or after the date of the first dose of double-blind study drug. Safety Set.
Arm/Group | Placebo | Lisdexamfetamine Dimesylate | Methylphenidate
Serious Adverse Events (participants affected / at risk) | 1/110 | 1/218 | 1/219
Other Adverse Events (participants affected / at risk) | 32/110 | 113/218 | 99/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=110) | Lisdexamfetamine Dimesylate (N=218) | Methylphenidate (N=219)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic episode (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=110) | Lisdexamfetamine Dimesylate (N=218) | Methylphenidate (N=219)
Weight decreased (Investigations) | 0 (0) | 23 (23) | 11 (11)
Headache (Nervous system disorders) | 9 (13) | 33 (45) | 35 (40)
Dizziness (Nervous system disorders) | 0 (0) | 12 (12) | 11 (11)
Irritability (General disorders) | 7 (7) | 11 (11) | 15 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 16 (18) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 11 (12) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 11 (11) | 8 (8)
Insomnia (Psychiatric disorders) | 3 (3) | 17 (17) | 17 (20)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 69 (74) | 51 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.